Effects of Early Community Services on Child and Family Development

ClinicalTrials.gov Identifier: NCT04019977

Last updated: July 18, 2023

## Statistical Analysis Plan

The principal independent variable will be MFC group (MFC participant/non-participant). The dependent variables of interest will be (a) infant emergency room use and overnight hospital stays; (b) family use of community resources and child care; (c) maternal wellbeing; and (d) quality of the home environment. We will also explore long-term differences between MFC and non-MFC participants in (a) rates of official investigations for child maltreatment and (b) two indicators of early educational achievement: kindergarten readiness scores and rates of kindergarten attendance.

A two-tailed intent-to-treat design analysis will include all randomly assigned families (regardless of actual intervention participation). Ordinary least squares regression models will be used to estimate impact of MFC on continuous and categorical outcomes. Poisson regression models will be used for count variables with skewed distribution. Covariates for all models will include the following: Medicaid status (yes/no) at birth and at 6 months, mother race/ethnicity (nonminority/minority), single parent household (yes/no), birth complications (yes/no) including maternal health conditions affecting the baby, infant injuries from birth trauma, and infant distress. Exploratory moderators will include infant birthweight, family Medicaid status, and mothers' adverse childhood experiences and adult attachment security. All results willbe analyzed at the .05 significance level.